CLINICAL TRIAL: NCT07229794
Title: Effect of Foot-ankle Exercise Using Elastic Band on Diabetic Foot Ulcer Incidence in Patient With Diabetes Neuropathy
Brief Title: Effect of Foot-ankle Exercise Using Elastic Band
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St Elisabeth School Health Science (Other)
Responsible Party: Principal Investigator, Maria Suryani, Principal investigator, St Elisabeth School Health Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Stikes Elisabeth11
Record Dates: First submitted 2025-09-22; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Foot Ulcer (DFU); Neuropathy (Disorder)
Keywords: diabetic foot ulcer; diabetes mellitus; foot ankle exercise; neuropathy diabetes
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- foot-ankle exercise group (Experimental): The group will receive usual care with additional food-ankle exercises using elastic band supervised by professional health care three times a week for twelve weeks. After twelve weeks period the patient will continue exercising for the completion of the study (9 month) by them self with the help of foot-ankle exercise video.
  Interventions: Other: foot-ankle exercise
- control group (No Intervention): Patient will receive usual care, with include pharmacological treatment and self care guidelines, which are maintained in both group

INTERVENTIONS:
Other: foot-ankle exercise — The exercise was done 3 times a week (15x/until they tired x 2set). The exercise used a elastic band with difference thickness (0,5 mm in 12 weeks and 0,65 mm in nine month)
  Arms: foot-ankle exercise group

SUMMARY:
The goal of this clinical trial is to learn if foot-ankle exercise can prevent diabetic foot ulcer incidence in patient with diabetes neuropathy. It will also learn about the effect of foot-ankle exercise on improvement of diabetes neuropathy severity, glycemic control, brain-derived neurotropic factor, walking speed, foot ankle range of motion, callus. The main questions it aims to answer are:

* Does foot-ankle exercise lower the number of diabetic ulcer incidence
* Does foot-ankle exercise lower the diabetes neuropathy severity
* Does foot-ankle exercise improve glycemic control
* Does foot-ankle exercise improve brain-derived neurotrophic factor
* Does foot-ankle exercise improve walking speed
* Does foot-ankle exercise improve foot ankle range of motion
* Does foot-ankle exercise lower the number of callus incidence

DETAILED DESCRIPTION:
Researchers will compare intervention group foot-ankle exercise used elastic band to a control group to see if foot-ankle exercise work to prevent diabetic foot ulcer incidence in patient with diabetes neuropathy

Participants will:

* Do foot-ankle exercise for three times a week with non-consecutive day for 1 year
* Report the incidence of callus and diabetic foot ulcer whenever they have

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* can walk minimal 10 meters
* neuropathy diabetic

Exclusion Criteria:

* stroke
* active ulcer
* fracture on foot area
* diabetic ulcer history

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
diabetic foot ulcer (DFU) incidence | for a year
  DFU, defined as a wound in the area below the ankle that reaches at least the epidermis and part of the dermis, as diagnosed by an internist

SECONDARY OUTCOMES:
diabetic neuropathy examination score | 0, 12 weeks, and a year
  The accumulation score of the result measurement consists of eight item, two testing muscle strength, one a tendon reflex, and five sensation. The min-max score is 0-16. The higher the score indicates the more severe the neuropathy. The score was determined by doing a physical examination.
control glyacemic | 0, 12 weeks, and a year
  HbA1c levels, which are the level of blood sugar control over a period of time. 3 months, measured by analyzing blood serum in a laboratory using the National Glycohemoglobin Standardization Program (NGSP).
brain derived neurotrophic factor | 0, 12 weeks, and a year
  BDNF levels, which are defined as biomolecular markers that can indicate the severity of diabetic neuropathy, as measured by analyzing blood serum using the ELIZA technique
walking speed | 0, 12 weeks, and a year
  Walking speed is the ratio between times measured while walking in second as fast as possible on a flat and flat trajectory at a certain distance. A track distance used in the study was 5 meter. The time of waking was measured using stopwatch
foot ankle range of motion | 0, 12 weeks, and a year
  ankle range of motion, which is the degree of joint movement in the feet during flexion, extension, inversion, and eversion, as measured using digital goniometry
callus insidence | 0, 12 weeks, and a year
  Callus is the thickness of the plantar skin area that can be determined by inspection
neuropathy symptom score | 0, 12 weeks, and a year
  The accumulation score of the result measurement consists of sixteen item about the symptom of neuropathy. The min-max score is 0-16. The more score indicates the more severe of neuropathy. The score was determined by interviewing the patient

CONTACTS AND LOCATIONS:
Overall Officials: maria suryani, Principal Investigator — stikes elisabeth
Locations (1):
- Elisabeth clinic, Semarang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT07229794/Prot_SAP_000.pdf